CLINICAL TRIAL: NCT04377230
Title: Impact of Biliopancreatic Limb Length of 60cm vs 100cm in Roux-en-Y Gastric Bypass on Bone Mineral Density 2 Years After Surgery
Brief Title: BP Limb Length of 60cm vs 100cm in Roux-en-Y Gastric Bypass
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital General Universitario Elche (Other)
Collaborators: Instituto de Seguridad Social del Estado de Mexico y Municipios (Other Government)
Responsible Party: Principal Investigator, Jaime Ruiz-Tovar, MD, PhD, Department of Surgery, Hospital General Universitario Elche
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Garcilaso-Mex 20-3
Record Dates: First submitted 2020-05-02; First posted 2020-05-06 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Osteopenia
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The radiologist evaluating bone mineral density will be blinded to the biliopancreatic limb length
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biliopancreatic limb 60cm (Experimental): Roux-en- Y gastric bypass will be performed with a biliopancreatic limb length of 60cm.
  Interventions: Procedure: biliopancreatic limb length of 60cm.
- Biliopancreatic limb 100cm (Active Comparator): Roux-en- Y gastric bypass will be performed with a biliopancreatic limb length of 100cm.
  Interventions: Procedure: biliopancreatic limb length of 100cm.

INTERVENTIONS:
Procedure: biliopancreatic limb length of 60cm. — Roux-en- Y gastric bypass will be performed with a biliopancreatic limb length of 60cm.
  Arms: Biliopancreatic limb 60cm
Procedure: biliopancreatic limb length of 100cm. — Roux-en- Y gastric bypass will be performed with a biliopancreatic limb length of 100cm.
  Arms: Biliopancreatic limb 100cm

SUMMARY:
Patients will be randomized into 2 groups:

* Group 60: Patients will undergo a Roux-en-Y gastric bypass with a Biliopancreatic limb length of 60cm
* Group 100: Patients will undergo a Roux-en-Y gastric bypass with a Biliopancreatic limb length of 100cm

Bone mineral density will be evaluated before surgery and 2 years after it.

DETAILED DESCRIPTION:
Patients will be randomized into 2 groups:

* Group 60: Patients will undergo a Roux-en-Y gastric bypass with a Biliopancreatic limb length of 60cm
* Group 100: Patients will undergo a Roux-en-Y gastric bypass with a Biliopancreatic limb length of 100cm Alimentary limb will be constant in both groups (150cm length)

Bone mineral density will be evaluated before surgery and 2 years after it, by means of X ray absorptiometry (DEXA). Changes in bone mineral density in lumbar column will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index >40 Kg/m2
* Body mass index >35 Kg/m2 associated to obesity related comorbidities

Exclusion Criteria:

* Bone pathologies
* Active neoplasms
* Disorders in calcium or vitamin D metabolism

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-05-07 (Estimated); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Bone mineral density | 2 years after surgery
  Bone mineral density will be evealuated by absorptiometry at the level of lumbar column

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Ruiz-Tovar, Principal Investigator — Garcilaso Clinic

IPD SHARING:
Plan to Share IPD: No